CLINICAL TRIAL: NCT07007767
Title: An Open-label, Single-arm, Exploratory Study of Sintilimab in Combination With Bevacizumab and Decitabine for the Treatment of Advanced pMMR/MSS Colorectal Cancer in Third-line or Later Settings
Brief Title: Exploring Sintilimab + Bevacizumab + Decitabine for Advanced pMMR/MSS Colorectal Cancer (After 2+ Prior Therapies）
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT-CRC-240601
Record Dates: First submitted 2025-05-15; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — sintilimab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sintilimab+bevacizumab+decitabine (Experimental): Subjects will receive Sintilimab (anti-PD-1 monoclonal antibody) in combination with Bevacizumab biosimilar（anti-VEGF monoclonal antibody) and Decitabine (hypomethylating agent) via intravenous infusion on a 3-week cycle (Q3W) until disease progression (PD), unacceptable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, loss to follow-up, death, or investigator-determined discontinuation criteria (whichever occurs first).
  The maximum treatment duration for Sintilimab is 24 months.
  Interventions: Drug: sintilimab; Drug: Bevacizumab Biosimilar; Drug: Decitabine

INTERVENTIONS:
Drug: sintilimab — Sintilimab (anti-PD-1 monoclonal antibody) Specification: 100 mg/10 mL (10 mg/mL concentrated solution)
  Administration:
  Dose: 200 mg (fixed dose) Route: Intravenous (IV) infusion over 30-60 minutes Schedule: Day 1 of each 21-day cycle (Q3W)
  Other Names: IBI308
Drug: Bevacizumab Biosimilar — Bevacizumab biosimilar (anti-VEGF monoclonal antibody) Specification: 100 mg/4 mL (25 mg/mL concentrated solution)
  Administration:
  Dose: 7.5 mg/kg (body weight-adjusted) Route: IV infusion Schedule: Day 1 of each 21-day cycle (Q3W)
  Other Names: IBI305
Drug: Decitabine — Decitabine (hypomethylating agent) Specification: 10 mg lyophilized powder per vial
  Administration:
  Dose: 10 mg/m²/day (body surface area-adjusted) Route: IV infusion over 1 hour Schedule: Days 1-5 of each 21-day cycle (Q3W)

SUMMARY:
This study investigates the efficacy and safety of sintilimab in combination with bevacizumab and decitabine for patients with advanced proficient mismatch repair/microsatellite stable (pMMR/MSS) colorectal cancer who have undergone ≥3 prior lines of systemic therapy.

Participants will receive intravenous infusions of sintilimab, bevacizumab, and decitabine in 3-week treatment cycles until disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, loss to follow-up, death, or investigator-determined discontinuation criteria (whichever occurs first). The maximum treatment duration for sintilimab is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to initiation of any trial-related procedures;
2. Age ≥18 years;
3. Histologically confirmed colorectal adenocarcinoma;
4. Microsatellite stable (MSS), microsatellite instability-low (MSI-L), or proficient mismatch repair (pMMR) status;
5. ECOG Performance Status (PS) score of 0-1;
6. Documented disease progression following standard second-line systemic therapy (prior exposure to irinotecan, oxaliplatin, or fluorouracil-based regimens, with or without targeted therapy [e.g., bevacizumab, cetuximab]);
7. Adequate organ and bone marrow function confirmed by laboratory parameters.
8. Anticipated survival exceeding 3 months.
9. For females of childbearing potential, a negative urine or serum pregnancy test must be confirmed within 3 days prior to the first dose of study drug (Cycle 1 Day 1). Serum pregnancy testing is required if urine results are inconclusive. Non-childbearing potential is defined as ≥1 year postmenopausal, surgically sterilized (bilateral oophorectomy or hysterectomy), or confirmed premature ovarian failure.
10. All subjects at risk of conception must employ highly effective contraception (failure rate <1% per year) throughout the treatment period and for 120 days after the last dose of study drug.
11. Subjects must consent to provide sufficient tumor tissue specimens for PD-L1 expression analysis, including archived samples (paraffin-embedded blocks or unstained sections meeting protocol-specified requirements). If archived tissue is unavailable, subjects must agree to undergo re-biopsy of the tumor lesion.

Exclusion Criteria:

1. Other malignancies diagnosed within the past 5 years, excluding radically resected basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
2. Microsatellite instability-high (MSI-H) or deficient DNA mismatch repair (dMMR).
3. Current participation in interventional clinical trials or administration of investigational drugs/devices within 4 weeks prior to the first dose.
4. Prior therapy with anti-PD-1/PD-L1/PD-L2 agents or drugs targeting stimulatory/coinhibitory T-cell receptors (e.g., CTLA-4, OX-40, CD137).
5. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Exemptions: Replacement therapy (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal/pituitary insufficiency).
6. Radiographic evidence of tumor invasion/encasement of major blood vessels or bleeding tendency assessed by investigators/radiologists.
7. Major surgery within 4 weeks prior to the first dose (excluding biopsy) or anticipated major surgery during the study period.
8. Non-healed wounds, ulcers, or fractures.
9. Minor surgical procedures (requiring local anesthesia, e.g., central venous catheterization) within 48 hours prior to the first dose.
10. Current or recent (within 10 days prior to the first dose) daily use of aspirin (>325 mg/day) or other NSAIDs with platelet-inhibiting effects.
11. Current or recent (within 10 days prior to the first dose) full-dose anticoagulants/thrombolytics (prophylactic low-dose anticoagulants permitted: ≤1 mg/day warfarin [INR ≤1.5], ≤12,000 U/day heparin, or ≤100 mg/day aspirin).
12. Inherited bleeding diathesis, coagulation disorders, or history of thrombosis.
13. History of allogeneic organ transplantation (excluding corneal transplants) or allogeneic hematopoietic stem cell transplantation.
14. Known hypersensitivity to sintilimab, bevacizumab, decitabine, or their excipients.
15. Inadequate recovery from prior intervention-related toxicities/complications (i.e., >Grade 1 or not returned to baseline, excluding fatigue/alopecia).
16. HIV infection (HIV 1/2 antibody-positive).
17. Untreated active hepatitis B (HBsAg-positive with HBV-DNA exceeding the upper limit of normal).
18. Pregnancy or lactation.
19. Severe or uncontrolled systemic diseases.
20. Any condition (medical, psychiatric, laboratory abnormality, or logistical) that, in the investigator's judgment, compromises patient safety, data integrity, or protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Investigator Assessment | every 12 weeks (±7 days) up to 2 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 is presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | every 12 weeks (±7 days) up to 2 years
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up. The OS is presented.
Overall Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator Assessment | every 12 weeks (±7 days) up to 2 years
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who experienced a CR or PR is presented.
Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator Assessment | every 12 weeks (±7 days) up to 2 years
  For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented.
Number of Participants Who Experienced an Adverse Event (AE) | Serious AEs: Up to 90 days after last dose of study treatment; Other AEs: Up to 30 days after last dose of study treatment
  An AE was defined as any untoward medical occurrence in a study participant administered study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who experienced an AE is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Ph.D., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be shared through presentations at international conferences or via publication in medical journals.
Supporting Information: Study Protocol, ICF
Time Frame: 2027/12/30
Access Criteria: After the research findings are publicly published